CLINICAL TRIAL: NCT05224999
Title: A Phase II Trial of Nivolumab for Recurrent/Metastatic Carcinosarcoma
Brief Title: Nivolumab for Recurrent/Metastatic Carcinosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-1104
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Recurrent/Metastatic Carcinosarcoma
Keywords: carcinosarcoma; nivolumab
MeSH Terms: conditions — Carcinosarcoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nivolumab (Experimental)
  Interventions: Drug: nivolumab

INTERVENTIONS:
Drug: nivolumab — nivolumab 3mg/kg (every 2 weeks)

SUMMARY:
Carcinosarcoma is a malignant neoplasm that is composed of both epithelial and mesenchymal elements and aggressive tumor that are staged as high-grade cancer in NCCN guideline. They are regarded as rare aggressive malignancies with a high potential to develop distant metastases and are associated with an overall poor survival. The aggressive nature of this malignancy coupled with a high relapse rate defines a poor clinical course for most patients. First line treatment of patients with advanced uterine carcinosarcoma with paclitaxel plus carboplatin achieved an objective response rate of 54% of patients. For this orphan tumor, carcinosarcoma, as these drugs would hypothetically act only on tissues with overexpression of PD-L1, they theoretically provide a more precise therapeutic effect on tumor cells with considerably less side effects. Therefore, the investigators suggest phase II trial of nivolumab for metastatic/recurred carcinosarcoma who have progressed after prior chemotherapy.

DETAILED DESCRIPTION:
Single center, prospective phase II trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed recurrent/metastatic carcinosarcoma
2. ECOG performance status of 0 to 1
3. ≥ 19 years of age
4. At least 1 prior chemotherapy
5. Patients who have at least 1 measurable disease per the RECIST Guideline Ver. 1.1 as confirmed by imaging within 28 days before randomization
6. Subjects who meet the following criteria:

   * Absolute neutrophil count (ANC) ≥ 1500 /µ
   * Platelet count ≥ 75,000/ µL
   * Serum creatinine < 1.5 x upper limit of normal (ULN)
   * AST (SGOT) and ALT (SGPT) < 3 x upper limit of normal (ULN) (If there is Liver Metastasis < 5 x upper limit of normal (ULN))
   * Total bilirubin < 1.5 x upper limit of normal (ULN)

Exclusion Criteria:

1. More than 4 prior cytotoxic agents
2. Prior treatment with systemic PD-L1-directed therapy
3. Patient who has had chemotherapy, radiotherapy, or biological therapy within 2 weeks prior to entering the study, or who has not recovered from the adverse events due to previous agents administered more than 2 weeks prior to study day
4. Subjects with symptomatic central nervous system (CNS) metastases who are neurologically unstable or have required increasing doses of steroids within the 2 weeks prior to study entry to manage CNS symptoms
5. Patients with multiple primary cancers (with the exception of completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, or superficial bladder cancer, or any other cancer that has not recurred for at least 3 years)
6. History of active non-infectious pneumonitis requiring treatment with steroids, or history or current signs of chronic interstitial lung disease
7. Known active infection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-11-13 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression free rate (PFR) at 6 months | at 6 months
  proportion of patients who did not progress and were alive at 24 weeks (RECIST version 1.1)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) by RECIST version 1.1 | 8 weeks
Progression-free survival (PFS) by RECIST version 1.1 | 8 weeks
Overall survival (OS) | 8 weeks
Time to progression (TPP) | 8 weeks
Drug toxicity and safety analysis by CTCAE Version 5 | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea